CLINICAL TRIAL: NCT03667196
Title: Evaluation of Effectiveness and Safety of Antegrade and Retrograde Approach of Percutaneous Coronary Intervention for Chronic Total Occlusions; Systemic Chronic Total Occlusion Revascularization Korea Research-Chronic Total Occlusion (STRIKE-CTO) Study
Brief Title: Evaluation of Effectiveness and Safety of Antegrade and Retrograde Approach of Percutaneous Coronary Intervention for Chronic Total Occlusions
Acronym: STRIKE-CTO
Status: Recruiting | Type: Observational
Sponsor: Seung-Whan Lee, M.D., Ph.D. (Other)
Collaborators: Abbott Medical Devices (Industry); Biotronik SE & Co. KG (Industry); Medtronic (Industry); Dio Medical (Unknown)
Responsible Party: Sponsor-Investigator, Seung-Whan Lee, M.D., Ph.D., M.D., Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV 2017-07
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational
  Interventions: Procedure: antegrade and retrograde approach

INTERVENTIONS:
Procedure: antegrade and retrograde approach — This study intends to identify and compare the clinical, anatomical and periprocedural factors of the patients who used only the antergrade approach and the patients who needed the retrograde approach among the patients with coronary CTO

SUMMARY:
Objective of this study is to 1) analyze the clinical, anatomical and periprocedural differences of patients who underwent a procedure related to coronary CTO through the antergrade approach and retrograde approach; 2) analyze the success rate of the procedures and the incidence and patterns of complications; 3) compare and analyze long-term performances after the successful procedure; and 4) identify the independent factors that require a retrograde approach and the prognostic factor regarding long-term performances after use of each approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged>=19
* Patients who have a CTO lesion in at least one or more epicardial coronary artery 2.5 mm in blood vessel diameter
* Patients who have symptoms of angina or objectively proven myocardial ischemia (asymptomatic myocardial ischemia, stable or unstable angina, non - -ST-segment elevation myocardial infarction)
* Patients who voluntarily agreed to the protocol and the clinical follow-up plan (or let their representative do this), and signed the informed consent form approved by the IRB of each study institute

Exclusion Criteria:

* Patients who are pregnant or lactating or have childbearing potential Patients in whom contrast medium and heparin are contraindicated or who are hypersensitive to them
* Patients in whom aspirin, clopidogrel, ticagrelor and prasugrel, cilostazol are contraindicated
* Patients scheduled to undergo a surgery, etc. that requires discontinuance of an antiplatelet drug within 12 months after participation in the study
* Acute ST elevation myocardial infarction at the time of hospitalization
* Terminally ill patients with their life expectancy < one year
* Patients who have serious diseases other than cardiac diseases that may affect limitation of residual life time or observation of the protocol (e.g. oxygen-independent chronic obstructive pulmonary disease, persisting hepatitis or serious hepatic insufficiency, severe renal disease, etc. Be left up to the discretion of the investigator.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will be determined after screening patients who undergo PCI for CTO lesions and completing the evaluation of all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 12-month after PCI
  Death
myocardial infarction | 12-month after PCI
  the periprocedural myocardial infarction under the SCAI definition or the non-lethal myocardial infarction during the follow-up observations
the complex endpoints of target vessel revascularization/reocclusion occurrence | 12-month after PCI
  including chronic total occlusion and angiostenosis

SECONDARY OUTCOMES:
Procedure success rate | every 1-year up-to 5-year
  A procedure success defined as the case where a final vessel diameter stenosis < 30% is achieved after the stent insertion
Myocardial infarction | every 1-year up-to 5-year
  Q-wave VS non-Q-wave, periprocedural myocardial infarction VS follow-up myocardial infarction (spontaneous myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (32):
- South Korea (32):
  - Hallym University Sacred Heart Hospital, Anyang
  - SoonChunHyang University Hospital Bucheon, Bucheon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Gangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - the Catholic University of Korea, Daejeon St. Mary'S Hospital, Daejeon
  - The Catholic University of Korea, ST. Vincent's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Myongji Hospital, Goyang-si
  - Hanyang University Medical Center, Guri-si
  - Gwangju Veterans Hospital, Korea Veterans Health Service, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Seoul national university Bundang hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - The Catholic University of Korea, Incheon ST. MARY'S Hospital, Incheon
  - Busan Veterans Hospital, Korea Veterans Health Service, Pusan
  - Dong-A University Hospital, Pusan
  - Gosin University Gospel Hospital, Pusan
  - Inje University Haeundae Paik Hospital, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Chungnam National University Sejong Hospital, Sejong
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong, Seoul
  - The Catholic University of Seoul St. Mary's Hospital, Seoul
  - Veterans Hospital Service Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided